CLINICAL TRIAL: NCT03516435
Title: Randomized,Single-Blind Controlled Trial
Brief Title: Efficacy of Different Electrical Stimulation Placement in Patients With Overactive Bladder Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Yeh, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS17150
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Overactive Bladder Syndrome
Keywords: Intravaginal electrical stimulation; Parasacral transcutaneous electrical stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parasacral transcutaneous ES (Experimental): 20min./session, 2 sessions/week ,12 sessions of Parasacral transcutaneous electrical stimulation.
  Interventions: Device: Parasacral transcutaneous electrical stimulation
- Intravaginal electrical stimulation (Active Comparator): 20min./session, 2 sessions/week ,12 sessions of Intravaginal electrical stimulation.
  Interventions: Device: Intravaginal electrical stimulation

INTERVENTIONS:
Device: Parasacral transcutaneous electrical stimulation — Asymmetrical biphasic square current pulse Frequency：10 Hz pulse width：1.0 ms Intensity：highest tolerable intensity(≦80 mA.) Parasacral transcutaneous electrical stimulation：Clinic using 2 superficial 3.5 cm electrodes placed on each side of S3 and S4.
  Arms: Parasacral transcutaneous ES
Device: Intravaginal electrical stimulation — Asymmetrical biphasic square current pulse Frequency：10 Hz pulse width：1.0 ms Intensity：highest tolerable intensity(≦80 mA.) Intravaginal electrical stimulation：The electrode plug for vaginal plug was cylinder-formed with ring-formed placed into vaginal.
  Arms: Intravaginal electrical stimulation

SUMMARY:
This experiment is expected to understand the benefits of different settings of electrical stimulation in the treatment of overactive bladder.

DETAILED DESCRIPTION:
This experiment is expected to understand the benefits of different settings of electrical stimulation in the treatment of overactive bladder.The study will adopt a longitudinal research design with randomized quasi-experimental trial.The patients will recruited and be randomly assigned to Group A (Parasacral transcutaneous electrical stimulation) or Group B (Intravaginal electrical stimulation). There will be 30 participants in each group. Data will be collected 2 times.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence due to detrusor overactivity
* No patients had been taking anticholinergics or tricyclic depressants and none had been treated by pelvic floor exercise, bladder training, or pelvic surgery before entry into the study.

Exclusion Criteria:

* stress incontinence
* urinary tract infection
* neurological disease
* genital prolapse higher than stage II on POP-Q system
* pregnancy
* diabetes mellitus
* a history of anti-incontinence surgery and/or prolapse repair
* pelvic tumors and previously treated with radiation therapy or antimuscarinic agents
* patients who were not cooperative
* electrical stimulation contraindications

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
3 Days Voiding diary | 3 days
  This chart is a record of your voiding and leakage or urine. Choose three (3) separate 24 hour periods to complete this record. Pick days which will be most convenient for you to measure every void.

SECONDARY OUTCOMES:
Overactive Bladder Symptom Score( OABSS） | 20 min
  This is a single symptom score that employs a self-report questionnaire to quantify OAB symptoms.Questionnaire has many items with the same minimum and maximum score.Four question items, daytime frequency, nocturia, urgency and urgency incontinence, were included in the questionnaire according to the definition of OAB.
minVisual analogue scale (VAS) for urgency | 10 min
  The Visual Analog or Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of urgency they experienced. This gives them the greatest freedom to choose their urgency intensity. It also gives the maximum opportunity for each respondent to express a personal response style. VAS data of this type is recorded as the number of millimeters from the left of the line with the range 0-100.
Pad test | 20min-1hr
  To measure leakage and may be performed in the specialist's office or at home. Pad testing can be done over a period of time as short as twenty minutes or up to one hour.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Gin-Den, PhD, Study Chair — Chung Shan Medical University; Chen Yi-Ching, MS, Study Director — Chung Shan Medical University; Chang Chia-Yun, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan